CLINICAL TRIAL: NCT06977503
Title: A Pilot Study Using a Cranial Electrotherapy Stimulation (CES) Device in Conjunction With Life Coaching to Alleviate Burnout Symptoms in HealthCare Workers (HCWs)
Brief Title: Electrotherapy Stimulation Together With Life Coaching for the Support of Burnout Symptoms in Healthcare Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: I-3956824; NCI-2025-03017 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3956824 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Researchers will be blinded with respect to subjects' study number, pre/post assessment data, and CES group (e.g., Group A versus Group B), the participants will remain blinded to which device they received (either sham or investigational device) throughout the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (Cranial Electrotherapy Stimulation (CES) + life coaching) (Experimental): During weeks 1-6, participants use the CES device QD over 1 hour 5 days per week for 6 weeks on study. Participants also participate in virtual group life coaching sessions and discussions and view video assignments 3 times during weeks 1, 3, and 6. At week 7 participants will return their devices and receive their second device . During weeks 8-13 participants cross-over and use the sham device QD over 1 hour 5 days per week for 6 weeks on study.
  Interventions: Other: Discussion; Behavioral: Health and Wellness Coach; Other: Informational Intervention; Other: Survey Administration
- Arm II (Sham device + life coaching sessions) (Sham Comparator): During weeks 1-6, participants use the sham device QD over 1 hour 5 days per week for 6 weeks on study. Participants also participate in virtual group life coaching sessions and discussions and view video assignments 3 times during weeks 1, 3, and 6. At week 7, participants return their device and receive their second device. During weeks 8-13, participants cross-over and use the CES device QD over 1 hour 5 days per week for 6 weeks on study.
  Interventions: Procedure: Cranial Electrical Stimulation (CES); Other: Discussion; Behavioral: Health and Wellness Coach; Other: Informational Intervention; Procedure: Sham Intervention; Other: Survey Administration

INTERVENTIONS:
Procedure: Cranial Electrical Stimulation (CES) — Use CES device
  Arms: Arm II (Sham device + life coaching sessions)
Other: Discussion — Participate in discussions
  Other Names: Discuss
Behavioral: Health and Wellness Coach — Undergo coaching sessions
Other: Informational Intervention — View video assignments
Procedure: Sham Intervention — Undergo sham intervention
  Other Names: Sham Comparator
  Arms: Arm II (Sham device + life coaching sessions)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the effect of life coaching together with Cranial Electrotherapy Stimulation (CES) as an intervention to decrease self-reported symptoms of burnout, moral distress, resilience, and employee retention in oncology healthcare workers. Burnout and moral distress are occupational hazards for oncology healthcare workers. Emotional exhaustion, depersonalization, and lack of personal accomplishment at work are symptoms of burnout. Moral distress may be defined as knowing the right thing to do but being unable to do so based upon internal or external constraints. The device is attached to the earlobes that uses cranial electrotherapy stimulation (CES) at a microcurrent to alleviate symptoms of anxiety, insomnia, pain, and possibly depression. Life coaching is partnering with clients in a thought-provoking and creative process that inspires them to maximize their personal and professional potential and can increase resiliency skills such as boundary setting and prioritizing, increases in self-compassion and self-care, and potentially indirectly positively impact patient care. Undergoing the use of CES via the CES device, coupled with life coaching, may help alleviate burnout symptoms and moral distress in oncology healthcare workers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of using Cranial Electrotherapy Stimulation (CES) with group life coaching sessions as an intervention to decrease healthcare worker self-reported symptoms of burnout and moral distress.

SECONDARY OBJECTIVE:

I. To determine the efficacy of using Cranial Electrotherapy Stimulation (CES) with group life coaching sessions as a supportive intervention to increase healthcare worker self-reported ratings of resilience, and employment retention (Organizational Wellbeing Assessment - Retention [OWA-R]).

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: During weeks 1-6, participants use the CES device once daily (QD) over 1 hour 5 days per week for 6 weeks on study. Participants also participate in virtual group life coaching sessions and discussions and view video assignments 3 times during weeks 1, 3, and 6. At week 7, participants exchange device for second device. During weeks 8-13, participants cross-over and use the sham device QD over 1 hour 5 days per week for 6 weeks on study.

ARM II: During weeks 1-6, participants use the sham device QD over 1 hour 5 days per week for 6 weeks on study. Participants also participate in virtual group life coaching sessions and discussions and view video assignments 3 times during weeks 1, 3, and 6. At week 7, participants exchange device for second device. During weeks 8-13, participants cross-over and use the CES device QD over 1 hour 5 days per week for 6 weeks on study.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 ≤ and ≤ 75 years old
* Patient-facing healthcare workers (e.g., medical doctor, advanced practice provider, nurse)
* Experiencing symptoms of burnout, as defined by a score of 1, 2, or 3 on question #2 of the Mini-Z II Survey
* Working on the Buffalo-Niagara Medical Campus (e.g. Roswell Park, Oishei Children's Hospital, Buffalo General, etc.)
* Ability to attend three (3) in-person appointments, one (1) hour in duration, at Roswell Park at week 1, week 6 and week 12 corresponding to the initial, midpoint, and final assessments
* Ability to use the CES daily for an hour each day

  * Although the device is water-resistant, participants must agree to not use the device in the bath or shower
* Ability to read and write in English
* Participant has access to a computer with internet access and an email address

  * Ability to attend three (3) virtual 60-minute group life coaching sessions, via Zoom
  * Ability to complete three (3) 10-15-minute pre-recorded video assignments, which will be distributed via email (each assignment will be due by the end of the week that they are distributed)
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Subjects who self-report as pregnant or nursing. Pregnancy be verified with a urine test for all persons of childbearing potential with a uterus
* Subjects with a self-reported history of the following: Meniere's disease, history of vertigo or prone to dizziness, seizure disorder, pacemaker / implantable cardioverter-defibrillator (automatic implantable cardioverter defibrillator [AICD]), cochlear implant, or any implanted electrical devices that cannot be shut off
* Inability to tolerate the required minimum stimulation amplitude (200 uA) during the initial device training at the baseline visit.
* Any self-reported medical or psychiatric condition which in the PI or study physician's opinion deems the participant an unsuitable candidate to participate in this trial.
* Unwilling or unable to follow protocol requirements

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Symptoms of burnout in healthcare workers (HCWs) | At baseline, 6 weeks, and 13 weeks
  Will be assessed using the Mini-Z Survey. Will be summarized by study arm and time-point (baseline, midpoint, and follow-up) using the appropriate descriptive statistics, and graphically using mean or dot plots. The Mini-Z scores will be modeled as a function of study arm, time-point, their two-way interaction, and random cohort and subject (nested within cohort) effects using linear mixed models (LMMs).
Symptoms of moral distress in HCWs | At baseline, 6 weeks, and 13 weeks
  Will be assessed using the Measure of Moral Distress for Healthcare Workers (MMDHW). Will be summarized by study arm and time-point (baseline, midpoint, and follow-up) using the appropriate descriptive statistics, and graphically using mean or dot plots. The MMDHW scores will be modeled as a function of study arm, time-point, their two-way interaction, and random cohort and subject (nested within cohort) effects using LMMs.

SECONDARY OUTCOMES:
Self-reported resilience in HCWs | At baseline, 6 weeks, and 13 weeks
  Measure of resilience will be assessed using the Brief Resilient Coping Scale. Will be summarized by study arm and time-point (baseline and follow-up) using the appropriate descriptive statistics, and graphically using mean or dot plots. Will be modeled as a function of study arm, time-point, their two-way interaction, and random cohort and subject (nested within cohort) effects using LMMs.
HCW self-reported probability of employment retention | At baseline, 6 weeks, and 13 weeks
  Likelihood of employment retention will be assessed using the Organizational Wellbeing Assessment - Retention. Will be summarized by study arm and time-point (baseline and follow-up) using the appropriate descriptive statistics, and graphically using mean or dot plots. Will be modeled as a function of study arm, time-point, their two-way interaction, and random cohort and subject (nested within cohort) effects using LMMs.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Gallagher, PsyD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States